CLINICAL TRIAL: NCT03289338
Title: Zoledronic Acid or Methylprednisolone in the Management of Active Charcot's Neuroarthropathy of Foot in Patients With Diabetes Mellitus: A Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Zoledronic Acid or Methylprednisolone for Active Charcot's Neuroarthropathy of Foot in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZoleMethCNO
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Charcot Arthropathy; Diabetes Complications
Keywords: Zoledronic acid; Methylprednisolone; Active Charcot's disease
MeSH Terms: conditions — Arthropathy, Neurogenic; Diabetes Complications | interventions — Zoledronic Acid; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Zoledronic acid (Experimental): Bisphosphonate Zoledronic acid
  Interventions: Drug: Zoledronic Acid
- Methylprednisolone (Active Comparator): Glucocorticoid Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Placebos (Placebo Comparator): Placebo normal saline
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid 5mg intravenous once a month for 3 months
  Other Names: Zoledronate
  Arms: Zoledronic acid
Drug: Methylprednisolone — Methylprednisolone 1gm intravenous once a month for 3 months
  Other Names: MPS
  Arms: Methylprednisolone
Drug: Placebos — Normal saline intravenous once a month for 3 months
  Other Names: NS
  Arms: Placebos

SUMMARY:
Charcot neuropathic osteoarthropathy (CNO) is a progressively destructive process resulting from significant peripheral neuropathy of almost any aetiology. Diabetes mellitus has emerged as the commonest cause of CNO.

The Charcot foot in diabetes poses many clinical challenges in its diagnosis and management. The lacuna primarily lies in delineation of its etio-pathogenesis and consequently in targeted treatment modalities. Although traditional approaches focus on neurotraumatic and neurovascular theories, these fail to explain all the features of CNO, hence, other hypotheses have been put forward.The current belief is that once the disease is triggered in a susceptible individual, it is mediated through a process of uncontrolled inflammation which, in turn, leads to osteolysis, fractures and joint destruction. Of these processes, the involvement of the receptor activator of nuclear factor- кB (RANK) ligand /RANK/osteoprotegerin (OPG) system in the process of acute CNO is particularly appealing and suggests new pharmacological approaches.

Standard modalities of treatment include offloading and casting. Although various trials have analysed the impact of medical agents including bisphosphonates, teriparatide and bone stimulation techniques, the results have been either inconclusive or not translated into clinical practice. Hence, there is no efficacious treatment of active CNO apart from the traditional offloading. In view of recent advances in understanding of the disease process, the target of intervention should, logically, be interruption of the inflammatory cascade and subsequent osteoclast resorption. Zoledronic acid is the most potent bisphosphonate that has been studied in clinical trials to date and has the distinctive profile of strong inhibitory activity on the enzyme farnesyl pyrophosphate synthase, essential for osteoclast function. Methylprednisolone conceivably has a potential benefit by offsetting the RANKL/OPG system involved. There have been conflicting reports with bisphophosphonates in active CNO and Zoledronic acid has been infrequently used despite being the most potent. Glucocorticoids including methylprednisolone have also not been systematically tried in this condition.

We hypothesise that targeting the inflammatory cascade with Methylprednisolone and osteoclast mediated damage by Zoledronic acid will address the basic etiopathogenesis of active CNO and may result in earlier resolution of the disease activity. The above mentioned hypothesis is hence, planned to be tested in a randomised, double-blind, placebo-controlled study.

DETAILED DESCRIPTION:
Charcot's neuroarthropathy has been identified since 1883, yet we have much to learn about the pathophysiology and evidence based treatment options. Active CNO is characterised by repetitive trauma leading to inflammation in an insensate foot. This includes polypeptide receptor activator of nuclear factor-kB ligand (RANKL) which triggers the synthesis of the nuclear transcription factor nuclear factor-kb (NF-kb), and this in turn stimulates the maturation of osteoclasts from osteoclast precursor cells. At the same time, NF-kb stimulates the production of the glycopeptide osteoprotegerin (OPG) from osteoblasts. This "decoy receptor" acts as an effective antagonist of RANKL . It has been suggested that this results in continual production of proinflammatory cytokines, RANKL, NF-kb, and osteoclasts, which in turn leads to continuing local osteolysis .This has adequately demonstrated by an increase in proinflammatory phenotypes of monocytes in those with active Charcot foot when compared with diabetic control subjects. Also osteoclasts generated in vitro in the presence of macrophage colony-stimulating factor and RANKL from patients with active CN have been shown to be more aggressive and exhibit an increase in their resorptive activity compared with control subjects. Motor neuropathy contributes to altered structure of the foot with resultant abnormal loading. Finally, it is possible that peptides like calcitonin gene-related peptide (CGRP) , which normally antagonizes the synthesis of RANKL, reduced due to neuropathy increase the RANKL expression. Diabetes may predispose to occurrence of CNO through a number of mechanisms. Apart from the presence of neuropathy and possible osteopenia, these include the effects of advanced glycation end products, reactive oxygen species, and oxidized lipids, which may all enhance the expression of RANKL in diabetes.

The average delay in the diagnosis of acute Charcot has been reported to be around 29 weeks. Common misdiagnoses include cellulitis, erysipelas, deep vein thrombosis (DVT), venous insufficiency, gout, pseudogout, acute inflammatory arthritis, fracture, sprain, tumor, septic arthritis, osteomyelitis, Sudeck's atrophy, and rheumatoid arthritis. Delay in prompt diagnosis and initiation of treatment results in progression of the pathology resulting in rigid osseous deformity of the foot increasing the risk of callus formation, ulceration, infection, and lower extremity amputation by 15- to 40-fold .With the propensity for misdiagnosis and high potential for progression to a rigid foot deformity, early recognition and prompt initiation of treatment is paramount.

Radiographs are the primary initial imaging method for evaluation of the foot in suspected CNO. However, they may initially be normal or show subtle fractures and dislocations. Magnetic resonance imaging (MRI) has a higher sensitivity that allows detection of subtle changes in the early stages of active CNO when X-rays could still be normal. MRI primarily images protons in fat and water and can depict anatomy and pathology in both soft tissue and bone in great detail because of its unique capability of differentiating tissues with high detail.

Treatment of CNO is aimed at offloading the foot, treating bone disease, and preventing further foot fractures. Because of the various etiologies of increased local bone resorption and/or secondary osteoporosis in patients with CNO and limited randomized placebo-controlled trials in this area, treatment guidelines are largely based on professional opinion rather than the highest level of clinical evidence. Hence, there remains a dearth of evidence based medical management for Charcot neuroarthropathy. Offloading at the acute active stage of the Charcot foot is the most important management strategy and could arrest the progression to deformity. Ideally, the foot should be immobilized in an irremovable total contact cast (TCC), which is initially replaced at 3 days, then checked each week. Edema reduction is often remarkable in the first few weeks of treatment. The cast should be changed frequently to avoid "pistoning" as the edema subsides.

However, It is important to take into consideration that TCC may actually have unfavorable consequences including unnatural stress patterns, increased instability, loss of muscle tone, proprioception and boe density.Also, they are not designed to affect the underlying physiological mechanisms that cause bone destruction.In this context, treatment by antiresorptive drugs emerges as an attractive option. Bone turnover in patients with active CNO is excessive, hence bisphosphonates, by inhibiting osteoclast mediated resorption, have an important role to play. However, there is little evidence to support their use at present.Both oral and intravenous bisphosphonates have been studied in the treatment of CNO in small randomized, double-blind, controlled trials or in retrospective controlled studies. Whatever the precise pathophysiological mechanism of CNO, bone resorption and osteoclastic hyperactivity is a major feature of the early acute stage of this condition and makes the use of bone-resorption-inhibiting agents such as bisphosphonates(BPs) a logical therapeutic approach. Theoretically, pharmacological treatment of CNO by BPs, which inhibit osteoclastic resorption and may have direct anti-inflammatory properties, might slow or even stop the bony destruction through its ability to cause macrophage apoptosis.

Selby et al first reported the use of a BP in the treatment of CNO. They administered 30 mg pamidronate i.v.,followed by five infusions of pamidronate 60 mg every 2 weeks for 12 weeks in six patients with diabetes and acute CNO. The treatment was associated with improvement in local pain and a significant reduction in the activity of the CNO as measured by the decrease in the temperature of the affected foot, from 3.4±0.7°C (mean±SE) to 1.0±0.5°C (p 0.05). There was also a significant reduction in bone turnover as judged by alkaline phosphatase (ALP) level, which fell by 25±3% compared with initial values (p<0.001). Stansberry et al in 1999 reported a decrease in peak cutaneous blood flow in response to the infusion of 90 mg pamidronate i.v. over 24 h in 20 patients with diabetes and CNO, suggesting a anti-inflammatory action of pamidronate. In 1999, Young reported anecdotally two cases of diabetic acute CNO treated with i.v. infusions of pamidronate associated with immobilisation. After 3 months, the clinical outcome was judged favourable with a reduction in clinical signs and an absence of deformity. Pakarinen et al. in 2002 retrospectively analysed clinical records and X-rays of 36 feet with CNO from 1994 to 2000. Eighteen patients received BPP treatment (pamidronate 30-60 mg i.v. once a week for 6 weeks) and no complications were registered. There was no statistically significant difference in casting time between patients who received (11 weeks) and patients who did not receive (13 weeks) pamidronate. In this series, pamidronate infusions were used for selected individuals without any striking benefits or disadvantages. Clinically, treatment with BP was associated with a more rapid decrease in skin temperature, but this effect was not sustained. Effect on the pain differed among studies, with one showing improvement but another showing none.Pakarinen et al tried Zoledronic acid and reported that it did not reduce the duration of immobilization. Rather there was an increase in total time for casting in subjects treated with Zoledronic acid.Similar observations about longer time of immobilization with the use of BPs was reported in the the recent multicentric observational audit of acute diabetic CNO in the UK.

Randomised trials looking into possible use of glucocorticoids in management of active CNO have not been undertaken, possibly because of only recent understanding of the role of acute inflammation triggering the osteolysis that characterizes CNO. Intravenous supra-pharmacological doses of corticosteroids have been used in various inflammatory and autoimmune conditions because they are cumulatively less toxic than sustained steroid treatment at lower quantitative dosage. Their action is supposed to be mediated through non-genomic actions within the cell. When corticosteroids are administered as pulses, an immediate profound anti-inflammatory effect is achieved, inflammatory damage is minimized , toxicity is low and there is no prolonged suppressive effect on the hypothalamic-pituitary axis. But there are no randomized trials looking into the efficacy and potential benefit of methylprednisolone in CNO as of date.

Hence this trial was designed to compare the therapeutic efficacy and profiles of two well known agents Zoledronic acid (antiresorptive) and Methylprednisolone (anti-inflammatory) in patients of diabetes mellitus with active CNO of foot.

ELIGIBILITY:
Inclusion Criteria:

Patients with Diabetes mellitus with active Charcot neuroarthropathy of foot as per following criteria:

Clinical criteria

1. Warm, swollen and erythematous foot
2. Skin temperature exceeding 2°C at the clinically suspected site of the affected foot compared with a similar site on the contralateral foot (infrared thermometer)

Radiologic criteria MRI suggestive of acute CNO-

1. Osteopenia
2. Joint subluxation
3. Normal or low normal marrow signal on T1 MRI
4. Bone marrow edema on T2W MRI
5. Microfractures
6. Cortical disruption
7. Several joints or bones
8. Preserved periarticular subcutaneous fat

Exclusion Criteria:

1. Infected foot ulcer
2. Osteoporosis at lumbar spine or hip
3. Gouty arthritis
4. Active peptic ulcer disease
5. Any prior long term steroid intake for asthma, SLE, RA or IBD in the last 3 months
6. eGFR 45 ml/min or less
7. Active dental caries
8. Active upper gastrointestinal disease
9. Uncorrected Vitamin D deficiency
10. Peripheral vascular disease (ABI 0.9 or less)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Time for resolution of active Charcot foot | 6 months

SECONDARY OUTCOMES:
Time for reduction in levels of inflammatory cytokines (>= 50%) | 6 months
Time for radiologic resolution/reduction on MRI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, DM, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Department of Endocrinology, PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Das L, Rastogi A, Jude EB, Prakash M, Dutta P, Bhansali A. Long-term foot outcomes following differential abatement of inflammation and osteoclastogenesis for active Charcot neuroarthropathy in diabetes mellitus. PLoS One. 2021 Nov 8;16(11):e0259224. doi: 10.1371/journal.pone.0259224. eCollection 2021. PMID 34748565